CLINICAL TRIAL: NCT01153698
Title: Observational Cohort Study to Evaluate the Safety and Efficacy of Switching From Lovenox (Enoxaparin) 40mg to Pradaxa (Dabigatran Etexilate) 220mg in Patients Undergoing Elective Total Hip or Knee Replacement Surgery
Brief Title: Pradaxa (Dabigatran Etexilate) VTE Prevention After Elective Total Hip or Knee Replacement Surgery
Status: Terminated | Type: Observational
Why Stopped: This trial was prematurely discontinued due to low enrolment.
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1160.118
Record Dates: First submitted 2010-06-29; First posted 2010-06-30 (Estimated); Results first posted 2013-01-04 (Estimated); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Venous Thromboembolism; Arthroplasty, Replacement
MeSH Terms: conditions — Venous Thromboembolism | interventions — Dabigatran

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- patients after hip or knee replacement
  Interventions: Drug: dabigatran

INTERVENTIONS:
Drug: dabigatran — anticoagulation

SUMMARY:
an open, prospective, observational study to collect data on safety (major bleeding events) and efficacy (symptomatic venous thromboembolism(VTE)) of a switch from Enoxaparin to dabigatran etexilate in patients with total knee replacement (TKR) and total hip replacement (THR)

ELIGIBILITY:
Inclusion criteria:

patients age 18 years or above undergoing elective total hip or knee replacement surgery

Exclusion criteria:

according to the label recommendation for Pradaxa 220 mg QD

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: specialist care
Sampling Method: Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2010-08; Primary Completion 2011-12-21 (Actual); Study Completion 2011-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (7):
- Austria (7):
  - 1160.118.43004 Boehringer Ingelheim Investigational Site, Braunau am Inn
  - 1160.118.43002 Boehringer Ingelheim Investigational Site, Ehebichl
  - 1160.118.43005 Boehringer Ingelheim Investigational Site, Graz
  - 1160.118.43016 Boehringer Ingelheim Investigational Site, Stolzalpe
  - 1160.118.43001 Boehringer Ingelheim Investigational Site, Vienna
  - 1160.118.43007 Boehringer Ingelheim Investigational Site, Vienna
  - 1160.118.43011 Boehringer Ingelheim Investigational Site, Vienna

REFERENCES:
- [Derived] Wurnig C, Clemens A, Rauscher H, Kleine E, Feuring M, Windhager R, Grohs J. Safety and efficacy of switching from low molecular weight heparin to dabigatran in patients undergoing elective total hip or knee replacement surgery. Thromb J. 2015 Nov 26;13:37. doi: 10.1186/s12959-015-0066-9. eCollection 2015. PMID 26612979

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 168 patients enrolled and treated. 161 of these patients received enoxaparin and switched to dabigatran etexilate (Pradaxa), 2 patients were only treated with dabigatran etexilate and 5 patients only received enoxaparin but did not switch to dabigatran etexilate.
Groups:
- All Patients: receiving at least one dose of enoxaparin 40mg or at least one dose of Pradaxa 220mg
Period: Overall Study
Arm/Group | All Patients
Started | 168 (Entered and treated.)
Completed | 139 (Completed Pradaxa treatment.)
Not Completed | 29
Not completed — Adverse Event | 12
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 2
Not completed — Switch to other anticoagulants | 4
Not completed — Other | 2
Not completed — Not treated with Pradaxa | 5

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 168
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.9 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96
  Male | 72

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Major Bleeding Events (MBE) During the Switch-/ Post-switch Treatment Period
Description: Major bleeding events were defined according to the modified McMaster criteria. The criteria for MBEs were: fatal; clinically overt associated with loss of haemoglobin >=20g/L in excess of what was expected; clinically overt leading to the transfusion of >=2 units packed cells or whole blood in excess of what was expected; symptomatic retroperitoneal, intracranial, intraocular or intraspinal; requiring treatment cessation; leading to re-operation.
Time Frame: From last enoxaparin administration until 24 hours after last Pradaxa intake( planned: knee replacement: Day 10 after surgery, hip replacement:Day 28-35 after surgery)
Population: Treated set (TS) reduced to patients with switch-/ post-switch period. TS includes all patients who received at least one dose of enoxaparin or at least one dose of Pradaxa.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Patients
Number analyzed (Participants) | 163
Percentage of participants | 0.61 [0.02 to 3.37]

2. Primary Outcome: Percentage of Patients With Symptomatic Venous Thromboembolic Events (sVTE) and All-cause Mortality Events During the Switch-/ Post-switch Treatment Period
Description: sVTE was defined as the composite of documented symptomatic proximal and distal deep vein thrombosis (DVT) and documented symptomatic non-fatal pulmonary embolism (PE).
Time Frame: From last enoxaparin administration until 24 hours after last Pradaxa intake (planned: knee replacement: Day 10 after surgery, hip replacement:Day 28-35 after surgery)
Population: TS reduced to patients with switch-/ post-switch period.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Patients
Number analyzed (Participants) | 163
Percentage of participants | 0 [0 to 2.24]

3. Secondary Outcome: Percentage of Patients With MBE During Total Treatment Period
Description: MBEs were defined according to the modified McMaster criteria. The criteria for MBEs were: fatal; clinically overt associated with loss of haemoglobin >=20g/L in excess of what was expected; clinically overt leading to the transfusion of >=2 units packed cells or whole blood in excess of what was expected; symptomatic retroperitoneal, intracranial, intraocular or intraspinal; requiring treatment cessation; leading to re-operation.
Time Frame: From first enoxaparin administration until 24 hours after last Pradaxa intake if switch to Pradaxa was performed or to 35 hours after last enoxaparin administration if no switch was performed
Population: TS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Patients
Number analyzed (Participants) | 168
Percentage of participants | 0.60 [0.02 to 3.27]

4. Secondary Outcome: Percentage of Patients With MBE During Pre-switch Treatment Period
Description: as for outcome 3
Time Frame: From first enoxaparin administration until last enoxaparin administration
Population: TS reduced to patients with pre-switch period.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Patients
Number analyzed (Participants) | 166
Percentage of participants | 0 [0 to 2.20]

5. Secondary Outcome: Percentage of Patients With sVTE and All-cause Mortality Events During Total Treatment Period
Description: sVTE was defined as the composite of documented symptomatic proximal and distal DVT and documented symptomatic non-fatal PE.
Time Frame: as for outcome 3
Population: TS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Patients
Number analyzed (Participants) | 168
Percentage of participants | 0 [0.00 to 2.17]

6. Secondary Outcome: Percentage of Patients With sVTE and All-cause Mortality Events During Pre-switch Treatment Period
Description: as for outcome 5
Time Frame: From first enoxaparin administration until last enoxaparin administration
Population: TS reduced to patients with pre-switch period.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Patients
Number analyzed (Participants) | 166
Percentage of participants | 0 [0.00 to 2.20]

7. Secondary Outcome: Percentage of Patients With sVTE and All-cause Mortality Events During Switch Treatment Period
Description: sVTE was defined as the composite of documented symptomatic proximal and distal DVT and documented symptomatic non-fatal PE.
  Symptomatic DVT is defined as clinically symptomatic venous thromboembolic event and symptomatic non-fatal PE is defined as symptomatic pulmonary embolism
Time Frame: From last enoxaparin administration until first Pradaxa intake
Population: TS reduced to patients with switch period.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Patients
Number analyzed (Participants) | 161
Percentage of participants | 0 [0.00 to 2.27]

8. Secondary Outcome: Percentage of Patients With Major Extra-surgical Site Bleedings During Total Treatment Period
Description: Major extra-surgical site bleedings include all major bleedings not occurred at surgical site
Time Frame: as for outcome 3
Population: TS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Patients
Number analyzed (Participants) | 168
Percentage of participants | 0 [0.00 to 2.17]

9. Secondary Outcome: Volume of Wound Drainage (Post-operative)
Description: Total volume of wound drainage is calculated as sum of volume drainage from end of surgery until first dose of Pradaxa plus volume drainage from first dose of Pradaxa and onwards.
Time Frame: From end of surgery (before first dosing) until 24 hours after last Pradaxa intake
Population: Treated Set (All patients with non-missing information for both, the volume drainage until first dose of Pradaxa and the volume drainage from first dose of Pradaxa and onwards).
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | All Patients
Number analyzed (Participants) | 129
ml | 462.1 (275.2)

10. Secondary Outcome: Percentage of Patients With Single Components of Composite of sVTE and All-cause Mortality Events During Total Treatment Period
Description: Total treatment period is defined from first enoxaparin administration to 24h after last Pradaxa intake or to 35h after last enoxaparin administration if no switch was performed.
Time Frame: From first enoxaparin administration until 24 hours after last Pradaxa intake ( planned: knee replacement: Day 10 after surgery, hip replacement:Day 28-35 after surgery)
Population: Treated Set
Measure: Number; unit: Number of participants
Arm/Group | All Patients
Number analyzed (Participants) | 168
Number of participants
  Documented symptomatic proximal DVT | 0
  Documented symptomatic distal DVT | 0
  Documented symptomatic non-fatal PE | 0
  All-cause mortality | 0

ADVERSE EVENTS:
Time Frame: Enoxaparin 40mg: From first enoxaparin administration until first Pradaxa intake (if switch was performed) otherwise until 35h after last Enoxaparin administration; Pradaxa 220mg: From first Pradaxa intake until 24h after last Pradaxa intake
Groups:
- Enoxaparin 40mg: All patients treated with enoxaparin
- Pradaxa 220mg: All patients treated with Pradaxa
Arm/Group | Enoxaparin 40mg | Pradaxa 220mg
Serious Adverse Events (participants affected / at risk) | 0/166 | 4/163
Other Adverse Events (participants affected / at risk) | 0/166 | 14/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Enoxaparin 40mg (N=166) | Pradaxa 220mg (N=163)
Pneumonia (Infections and infestations) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Device dislocation (General disorders) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Enoxaparin 40mg (N=166) | Pradaxa 220mg (N=163)
Seroma (Injury, poisoning and procedural complications) | 0 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.